CLINICAL TRIAL: NCT06390163
Title: Investigation the Effects of Sensory-Motor Integration Training on Cognitive Functions, Balance and Gait in Patients with Idiopathic Parkinson's Disease
Brief Title: Effects of Sensory-Motor Integration Training in Patients with Idiopathic Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Seckinogullari Korkusuz, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-23038
Record Dates: First submitted 2024-03-01; First posted 2024-04-30 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Balance; Gait; Cognitive Function; Sensory-perception-motor training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sensory-motor Integration Training (Experimental): Patients in the study group will receive sensory-motor integration training for 60 minutes, 3 days a week for 8 weeks, in addition to their routine lives.
  Interventions: Other: Sensory-Motor Integration Training
- Standart Care (No Intervention): Patients in the control group will be asked to continue their routine lives and return for evaluation after 8 weeks. Individuals in the control group will be followed without any additional treatment or advice.

INTERVENTIONS:
Other: Sensory-Motor Integration Training — An exercise chain consisting of motor tasks, sensory stimuli and cognitive tasks will be created. Each session will include at least 3 motor tasks, 3 sensory stimuli and 3 cognitive tasks selected according to the patient's condition.
  Arms: Sensory-motor Integration Training

SUMMARY:
The goal of this single blind randomized controlled trial is to investigate the effect of sensory-motor integration training on cognitive functions, balance and gait in patients with Parkinson Disease?

The main questions it aims to answer are:

* Does sensory-motor integration training have an effect on balance in patients with Parkinson Disease?
* Does sensory-motor integration training have an effect on cognitive functions in patients with Parkinson Disease?
* Does sensory-motor integration training have an effect on gait in patients with Parkinson Disease? Patients in the control group will be asked to continue their routine lives and return for evaluation after 8 weeks. Individuals in the control group will be followed without any additional treatment or advice. Patients in the study group will receivesensory-motor integration training for 60 minutes, 3 days a week for 8 weeks, in addition to their routine lives. No additional recommendations will be given to individuals in either group.

DETAILED DESCRIPTION:
40 patients will be included in the study. Patients who agree to participate in the study will be divided into two groups, study and control groups, by using a table of random numbers, ensuring that there are equal numbers of patients in each group. Demographic and clinical information of all patients participating in the study will be recorded. Montreal Cognitive Assessment Test and Modified Hoehn Yahr Staging Scale scores of all participants will be recorded by the neurologist and eligible patients will be included in the study. Evaluations to be applied to the groups within the scope of the study: Unified Parkinson Disease Rating Scale Part 3 , Static posturography measurement, Functional Reaching Test , Dynamic Gait Index , Rapid Mild Cognitive Impairment Screening, Stroop Test, Symbol Digit Modalities Test , Clock Drawing Test. Assessments will be made during the patients on period (approximately 60 minutes after medication intake). On the first day of the study, demographic information will be recorded in both groups and the patients participating in the study will be randomized. After randomization, patients in the control group will be asked to continue their routine lives and return for evaluation after 8 weeks. Individuals in the control group will be followed without any additional treatment or advice. Patients in the study group will receive sensory-perceptual-motor training for 60 minutes, 3 days a week for 8 weeks, in addition to their routine lives. No additional recommendations will be given to individuals in either group. Patients will be excluded from the study if they participate in any physiotherapy and rehabilitation program during the study. Patients in both groups will be evaluated a total of 3 times: at the beginning of the study, at the end of the study (at week 8), and 4 weeks after the end of the study (at week 12).

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with idiopathic Parkinson's disease
* Being between the ages of 45-75
* Being between stage 2-3 according to the Modified Hoehn-Yahr Staging Scale
* Having a score > 21 on the Montreal Cognitive Assessment Scale
* Being literate in Turkish
* No drug or dose changes throughout the study.
* Not having participated in any physiotherapy or rehabilitation program in the last 6 months.
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of other neurological diseases
* Presence of vision problems (that cannot be compensated with the correct lens) or vestibular disorders that may affect balance, other than symptoms related to Parkinson's disease.
* Serious comorbidities that affect balance and gait or cannot be controlled with life-threatening medication (Diabetes, Hypertension, Cardiopulmonary diseases)
* Long-term corticosteroid use
* Presence of orthopedic and systemic diseases that may affect participation in exercise

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Static Posturography | Baseline, week 8 and week 12
  It measures postural stability while standing statically and dynamically. The device has a computer-connected force platform that measures the vertical forces applied on the patients' feet (center of pressure/COG) to measure the position of the center of gravity and postural control.
Modified Dynamic Gait Index | Baseline, week 8 and week 12
  Index is used to evaluate and document the ability to respond to changing task demands during gait. An increase in the score indicates that the patient's walking ability is better.
Functional Reach Test | Baseline, week 8 and week 12
  It is used to evaluate dynamic balance and anteroposterior stability. In the standing position, the arm is lifted 90° upwards and stretched forward as much as possible, without losing contact with the feet. Initially, the projection of the acromion and the 3rd metacarpal bone on the wall is marked. At the final point reached after reaching forward, the projection of the 3rd metacarpal bone on the wall is marked and the difference is calculated. In elderly individuals, there is a risk of falling if the reach distance is less than 25.4 cm, and there is a risk of serious falling if it is less than 15 cm.
Quick Mild Cognitive Impairment Screen | Baseline, week 8 and week 12
  It consists of 6 subtests: orientation, registration, clock drawing, delayed recall, verbal fluency and logical memory. This has a high degree of sensitivity in detecting cognitive impairment. It is also quick to apply, taking 3 to 5 minutes. There are cutoff points that are adjusted for factors such as age and education level. The total score is 100, and a score below 62 points indicates cognitive impairment.
Symbol Digit Modalities Test | Baseline, week 8 and week 12
  It is a test frequently used in clinics because it evaluates attention, visuo-spatial information processing speed and working memory. Test is based on matching meaningless geometric shapes with certain numbers. The first 10 symbols are considered trials. Then the test starts and the person gets points for the correct marking he makes within 90 seconds. The maximum score is 60. Turkish Standardization of the test battery containing the relevant test was made and permission was obtained from the relevant authors
Stroop Test | Baseline, week 8 and week 12
  The Stroop Test, which also measures the ability to change perceptual setup and response under disruptive influence, information processing speed and attention (especially selective attention).Increasing time and error indicates lower cognitive level.
Clock Drawing Test | Baseline, week 8 and week 12
  Clock drawing test is an easy, quickly applicable, paper-and-pencil test with high validity and reliability used to evaluate visual-motor functions, planning, sequencing and abstract thinking skills. The Shulmann method will be used for scoring and this method evaluates out of a total of 5 points. An increase in the score indicates a better cognitive level.
Movement Disorders Society Unified Parkinson's Disease Rating Scale - Part 3 | Baseline, week 8 and week 12
  It is the revised form developed in 1980, by the Movement Disorders Association in 2008. It is a revised version that will eliminate the uncertainties present in scale and include current scientific developments. The number of questions, which was 42 in scale, was increased to 50 , and questions with yes/no options were removed because they caused structural inconsistency, and all questions were scored between 0 and 4. In our study, only the 3rd Part, which includes the Motor examination, will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Fil Balkan, Assoc.Prof, Study Director — Hacettepe University; Süleyman Korkusuz, PhD, Study Chair — Atılım University; Ayşenur Özcan, MSc, Study Chair — Çankırı Karatekin University; Gül Yalçın Çakmaklı, Assoc.Prof., Study Chair — Hacettepe University; Öznur Yiğit, Assisst.Prof, Study Chair — Hacettepe University; Bülent Elibol, Prof.Dr., Study Chair — Hacettepe University; Büşra Seçkinoğulları Korkusuz, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gandolfi M, Munari D, Geroin C, Gajofatto A, Benedetti MD, Midiri A, Carla F, Picelli A, Waldner A, Smania N. Sensory integration balance training in patients with multiple sclerosis: A randomized, controlled trial. Mult Scler. 2015 Oct;21(11):1453-62. doi: 10.1177/1352458514562438. Epub 2015 Jan 12. PMID 25583852
- [Background] Taghizadeh G, Azad A, Kashefi S, Fallah S, Daneshjoo F. The effect of sensory-motor training on hand and upper extremity sensory and motor function in patients with idiopathic Parkinson disease. J Hand Ther. 2018 Oct-Dec;31(4):486-493. doi: 10.1016/j.jht.2017.08.001. Epub 2017 Nov 14. PMID 29150384